CLINICAL TRIAL: NCT04439591
Title: Group-based Brain-computer Interface (BCI) Cognitive Training in Healthy Older Adults: An Evaluation of Programme Implementation and Effectiveness in Neighborhood Community Centers
Brief Title: Evaluation of Implementation and Effectiveness of Computerised Brain Training for Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geriatric Education and Research Institute (Other Government)
Collaborators: Neeuro Pte Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2017/00611
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Cognition
Keywords: Computerised cognitive training; Healthy older adults

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention group undergoes computerised brain training programme first.
  Interventions: Other: Computerised cognitive training
- Control group (Other): Waitlist control group: control group undergoes programme after intervention group has completed it in a crossover design.
  Interventions: Other: Computerised cognitive training

INTERVENTIONS:
Other: Computerised cognitive training — A 12-week bi-weekly group-based computerised cognitive training programme conducted in community centres

SUMMARY:
This study aims to evaluate the implementation and effectiveness of a group-based brain-computer interface cognitive training among community dwelling older adults in Singapore. A 12-week bi-weekly programme was conducted in community centres. During these sessions, participants played games targeting cognitive domains such as attention, memory, and decision making, using a mobile application (Memorie). Selected games were paired with an electroencephalography headset (Senzeband) which quantified participants' attention level into scores that affected the participants' in-game avatar control or game performance. Each participant paid a subsidized fee of SGD$20 for the programme.

DETAILED DESCRIPTION:
There has been emerging interest in research to help older adults maintain cognitive and physical function in old age. There has been evidence that cognitive training can help improve targeted cognitive domains in both typically and atypically aging older people. Cognitive training typically involves structured, frequent and repeated engagement in standardized cognitively demanding tasks targeting specific cognitive domains. There are several potential mechanisms underlying cognitive benefits of cognitive training. As the brain has neural plasticity (which is the lifelong ability for physical and functional change in response to sensing, perceiving and learning), engaging in mentally stimulating activities may stimulate neuroplasticity and thereby increase cognitive reserve. In fact, animal studies have shown that cognitive stimulation can result in molecular, synaptic and neural alterations in the brain. Studies in humans also showed that intervention studies incorporating brain training have reported increased serum levels of brain derived neurotropic factor, a factor that plays an important role in memory processing. Brain imaging studies showed changes in activity in certain brain regions while performing specific tasks, along with long-term global changes following cognitive training. Over the last five years, there has been an increase in research about the effectiveness of CCT. According to a systematic review of the clinical significance of commercially available CCT in preventing cognitive decline in 2016, there have been 18 commercial brain training programs for older people. According to a meta-analysis of 52 studies using commercial CCT programs in 4885 participants, CCT is modestly effective at improving cognitive performance in cognitively healthy older adults, but efficacy varies across cognitive domains and is largely determined by design choices. Unsupervised at-home training and training more than three times per week are specifically ineffective. Small to moderate effect sizes were found for nonverbal memory, g = 0.24 (95% CI 0.09 to 0.38), verbal memory, g = 0.08 (95% CI 0.01 to 0.15), working memory (WM), g = 0.22 (95% CI 0.09 to 0.35), processing speed, g =0.31 (95% CI 0.11 to 0.50), visuospatial skills, g = 0.30 (95% CI 0.07 to 0.54), and no significant effect was found for executive function and attention. In Singapore, two previous randomized control trials also reported the benefits of CCT on improved overall RBANS score in healthy older adults, but the efficacy on targeted cognitive domains (memory, visuospatial, attention) was not consistent among these two studies.

Cognition has a close association with gait and balance. Cognitive impairments, specifically deficits in executive function, have been associated with increased risk of falls, abnormal gait, and other mobility tasks. Gait variability in older people is associated with atrophy in brain regions related to attention function. Global cognitive function, verbal memory, and executive function can predict longitudinal gait speed decline. There has been evidence that cognitive intervention may not only improve various cognitive domains but also improve physical function. As there has been no previously published review on the topic, the researchers conduct a literature search via MEDLINE (to May 2017). Keywords used for searching included "computerized cognitive training", "gait" and "balance". The articles attained by this search method were screened by title and three relevant original studies were retrieved. All of these studies were conducted in the United States. These studies suggested that CCT may improve gait speed and balance in American older people, especially in those with sedentary lifestyle. One such CCT programme in Singapore was developed by Neeuro together with A*STAR and was made commercially available since 2016. Since then, it has been showcased at various events, such as the Silver IT Fest and NextStop Seminar organised by the Future Ready Committee. To date, there has been no assessment on the effectiveness of CCT in cognition, gait and function in the older people in Singapore hence this study will focus on evaluating these parameters. Results from this study may contribute to evidence in the local context.

ELIGIBILITY:
Inclusion Criteria:

* Above or equal to 55 years old
* Sedentary lifestyle (exercise less than or equal to once week)
* Literate in English/Chinese
* Able to travel to study site independently

Exclusion Criteria:

* Had significant cognitive impairment (Mini Mental State Examination score <=23) or presence of known neuropsychiatric disorders
* Geriatric Depression Scale >9
* Presence of a severe walking or balance impairments
* Previously completed a cognitive training program within the last year
* Color-blindness
* Plans to begin a balance program during the study period
* Self-reported presence of vertigo
* Visual acuity of less than 20/80
* Currently using psychotropic medications

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-11-09 (Actual); Study Completion 2018-11-09 (Actual)

PRIMARY OUTCOMES:
Change in cognition from baseline at 12 weeks | Baseline and 12 weeks
  Repeated Battery for the Assessment of Neuropsychological Status (RBANS). The maximum score that an individual can get is 160, and higher scores indicate better performance. The tests consists of 12 subtests grouped into 5 domains of cognition.
Change in attention from baseline at 12 weeks | Baseline and 12 weeks
  Colour Trails Test. Time taken to complete the actual trial was recorded, along with the number of near-misses, prompts, number sequence errors, and color sequence errors.

SECONDARY OUTCOMES:
Change in balance from baseline at 12 weeks | Baseline and 12 weeks
  Berg Balance Scale (BBS). BBS provides a measure of balance via performance on 14 functional tasks. Performance for each task was scored independently using a 0 - 4 scale, with higher scores reflecting higher functioning and better balance. Individual task scores were summed to derive a composite score for analyses.
Change in walking gait from baseline at 12 weeks | Baseline and 12 weeks
  Portable gait analysis system (GAITRite). The GAITRite measures how a person walks. It measures gait patterns for both time (temporal) and space (spatial) through pressure sensors in the mat. The software changes the information into foot placement patterns and overall gait patterns.

CONTACTS AND LOCATIONS:
Overall Officials: Shiou Liang Wee, PhD, Principal Investigator — Geriatric Education and Research Institute
Locations (1):
- Geriatric Education and Research Institute, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Due to confidentiality issues, IPD will not be published. However, de-identified data will be made available upon request.

REFERENCES:
- [Background] Shah TM, Weinborn M, Verdile G, Sohrabi HR, Martins RN. Enhancing Cognitive Functioning in Healthly Older Adults: a Systematic Review of the Clinical Significance of Commercially Available Computerized Cognitive Training in Preventing Cognitive Decline. Neuropsychol Rev. 2017 Mar;27(1):62-80. doi: 10.1007/s11065-016-9338-9. Epub 2017 Jan 14. PMID 28092015
- [Background] Bahar-Fuchs A, Clare L, Woods B. Cognitive training and cognitive rehabilitation for mild to moderate Alzheimer's disease and vascular dementia. Cochrane Database Syst Rev. 2013 Jun 5;2013(6):CD003260. doi: 10.1002/14651858.CD003260.pub2. PMID 23740535
- [Background] Raz N, Lindenberger U. Life-span plasticity of the brain and cognition: from questions to evidence and back. Neurosci Biobehav Rev. 2013 Nov;37(9 Pt B):2195-200. doi: 10.1016/j.neubiorev.2013.10.003. Epub 2013 Oct 15. PMID 24140011
- [Background] Buonomano DV, Merzenich MM. Cortical plasticity: from synapses to maps. Annu Rev Neurosci. 1998;21:149-86. doi: 10.1146/annurev.neuro.21.1.149. PMID 9530495
- [Background] Anderson-Hanley C, Arciero PJ, Brickman AM, Nimon JP, Okuma N, Westen SC, Merz ME, Pence BD, Woods JA, Kramer AF, Zimmerman EA. Exergaming and older adult cognition: a cluster randomized clinical trial. Am J Prev Med. 2012 Feb;42(2):109-19. doi: 10.1016/j.amepre.2011.10.016. PMID 22261206
- [Background] Vinogradov S, Fisher M, Holland C, Shelly W, Wolkowitz O, Mellon SH. Is serum brain-derived neurotrophic factor a biomarker for cognitive enhancement in schizophrenia? Biol Psychiatry. 2009 Sep 15;66(6):549-53. doi: 10.1016/j.biopsych.2009.02.017. Epub 2009 Apr 15. PMID 19368899
- [Background] Buschert V, Bokde AL, Hampel H. Cognitive intervention in Alzheimer disease. Nat Rev Neurol. 2010 Sep;6(9):508-17. doi: 10.1038/nrneurol.2010.113. Epub 2010 Aug 17. PMID 20717104
- [Background] Lampit A, Hallock H, Valenzuela M. Computerized cognitive training in cognitively healthy older adults: a systematic review and meta-analysis of effect modifiers. PLoS Med. 2014 Nov 18;11(11):e1001756. doi: 10.1371/journal.pmed.1001756. eCollection 2014 Nov. PMID 25405755
- [Background] Lee TS, Goh SJ, Quek SY, Phillips R, Guan C, Cheung YB, Feng L, Teng SS, Wang CC, Chin ZY, Zhang H, Ng TP, Lee J, Keefe R, Krishnan KR. A brain-computer interface based cognitive training system for healthy elderly: a randomized control pilot study for usability and preliminary efficacy. PLoS One. 2013 Nov 18;8(11):e79419. doi: 10.1371/journal.pone.0079419. eCollection 2013. PMID 24260218
- [Background] Lee TS, Quek SY, Goh SJ, Phillips R, Guan C, Cheung YB, Feng L, Wang CC, Chin ZY, Zhang H, Lee J, Ng TP, Krishnan KR. A pilot randomized controlled trial using EEG-based brain-computer interface training for a Chinese-speaking group of healthy elderly. Clin Interv Aging. 2015 Jan 9;10:217-27. doi: 10.2147/CIA.S73955. eCollection 2015. PMID 25624754
- [Background] Muir SW, Gopaul K, Montero Odasso MM. The role of cognitive impairment in fall risk among older adults: a systematic review and meta-analysis. Age Ageing. 2012 May;41(3):299-308. doi: 10.1093/ageing/afs012. Epub 2012 Feb 27. PMID 22374645
- [Background] Holtzer R, Friedman R, Lipton RB, Katz M, Xue X, Verghese J. The relationship between specific cognitive functions and falls in aging. Neuropsychology. 2007 Sep;21(5):540-8. doi: 10.1037/0894-4105.21.5.540. PMID 17784802
- [Background] Kearney FC, Harwood RH, Gladman JR, Lincoln N, Masud T. The relationship between executive function and falls and gait abnormalities in older adults: a systematic review. Dement Geriatr Cogn Disord. 2013;36(1-2):20-35. doi: 10.1159/000350031. Epub 2013 May 23. PMID 23712088
- [Background] Persad CC, Jones JL, Ashton-Miller JA, Alexander NB, Giordani B. Executive function and gait in older adults with cognitive impairment. J Gerontol A Biol Sci Med Sci. 2008 Dec;63(12):1350-5. doi: 10.1093/gerona/63.12.1350. PMID 19126848
- [Background] Rosano C, Brach J, Studenski S, Longstreth WT Jr, Newman AB. Gait variability is associated with subclinical brain vascular abnormalities in high-functioning older adults. Neuroepidemiology. 2007;29(3-4):193-200. doi: 10.1159/000111582. Epub 2007 Nov 27. PMID 18043004
- [Background] Watson NL, Rosano C, Boudreau RM, Simonsick EM, Ferrucci L, Sutton-Tyrrell K, Hardy SE, Atkinson HH, Yaffe K, Satterfield S, Harris TB, Newman AB; Health ABC Study. Executive function, memory, and gait speed decline in well-functioning older adults. J Gerontol A Biol Sci Med Sci. 2010 Oct;65(10):1093-100. doi: 10.1093/gerona/glq111. Epub 2010 Jun 25. PMID 20581339
- [Background] Smith-Ray RL, Hughes SL, Prohaska TR, Little DM, Jurivich DA, Hedeker D. Impact of Cognitive Training on Balance and Gait in Older Adults. J Gerontol B Psychol Sci Soc Sci. 2015 May;70(3):357-66. doi: 10.1093/geronb/gbt097. Epub 2013 Nov 5. PMID 24192586
- [Background] Verghese J, Mahoney J, Ambrose AF, Wang C, Holtzer R. Effect of cognitive remediation on gait in sedentary seniors. J Gerontol A Biol Sci Med Sci. 2010 Dec;65(12):1338-43. doi: 10.1093/gerona/glq127. Epub 2010 Jul 19. PMID 20643703
- [Background] Blackwood J, Shubert T, Fogarty K, Chase C. The Impact of a Home-Based Computerized Cognitive Training Intervention on Fall Risk Measure Performance in Community Dwelling Older Adults, a Pilot Study. J Nutr Health Aging. 2016 Feb;20(2):138-45. doi: 10.1007/s12603-015-0598-5. PMID 26812509
- [Background] Billingham SA, Whitehead AL, Julious SA. An audit of sample sizes for pilot and feasibility trials being undertaken in the United Kingdom registered in the United Kingdom Clinical Research Network database. BMC Med Res Methodol. 2013 Aug 20;13:104. doi: 10.1186/1471-2288-13-104. PMID 23961782
- [Derived] Yeo PS, Nguyen TN, Ng MPE, Choo RWM, Yap PLK, Ng TP, Wee SL. Evaluation of the Implementation and Effectiveness of Community-Based Brain-Computer Interface Cognitive Group Training in Healthy Community-Dwelling Older Adults: Randomized Controlled Implementation Trial. JMIR Form Res. 2021 Apr 27;5(4):e25462. doi: 10.2196/25462. PMID 33904819